CLINICAL TRIAL: NCT06250244
Title: A Dosimetry Study and Dose-escalation and of [177Lu]Lu-LNC1011 in Metastatic Castration-Resistant Prostate Cancer Patients
Brief Title: 177Lu-LNC1011 in Patients with Metastatic Castration-resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NM-PSMA1011
Record Dates: First submitted 2024-01-10; First posted 2024-02-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: PSMA; 177Lu; mCRPC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LNC1011 Dose escalation (Experimental): Patients received a single dose of 1.85 GBq (50 mCi) of 177Lu-LNC1011 via intravenous injection, followed by monitoring at 3, 24, 48, 72, and 168 hours post-injection. Subsequent cohorts received a dose escalation of 0.925 GBq from the previous cohort.
  Interventions: Drug: 177Lu-LNC1011

INTERVENTIONS:
Drug: 177Lu-LNC1011 — [177Lu]Lu-LNC1011 is a novel long-circulating PSMA therapeutic probe.

SUMMARY:
This study employed an open-label, non-randomized design, representing the first human trial of its kind. It utilized a standard 3+3 dose-escalation approach, focusing on patients with metastatic castration-resistant prostate cancer, initiating treatment at a dose of 1.85 GBq over a 6-week period. Subsequent cohorts underwent sequential 50% dose escalations until the observation of dose-limiting toxicity (DLT).

DETAILED DESCRIPTION:
[177Lu]Lu-LNC1011 is a novel long-circulating PSMA therapeutic probe. This study represents the first human investigation, aiming to explore its maximum tolerated dose (MTD), safety, dosimetry, and initial treatment efficacy in patients with metastatic castration-resistant prostate cancer (mCRPC).This study employed an open-label, non-randomized design, representing the first human trial of its kind. It utilized a standard 3+3 dose-escalation approach, focusing on patients with metastatic castration-resistant prostate cancer, initiating treatment at a dose of 1.85 GBq over a 6-week period. Subsequent cohorts received a dose escalation of 0.925 GBq from the previous cohort.

ELIGIBILITY:
Inclusion Criteria:

* progressive metastatic castration-resistant prostate cancer
* tumors with high PSMA expression confirmed on 68Ga-PSMA PET/CT PSMA expression confirmed on 68Ga-PSMA PET/CT

Exclusion Criteria:

* a serum creatinine level of more than 150 μmol per liter
* a hemoglobin level of less than 10.0 g/dl
* a white-cell count of less than 4.0× 109/L
* a platelet count of less than 100 × 109/L
* a total bilirubin level of more than 3 times the upper limit of the normal range
* a serum albumin level of more than 3.0 g per deciliter
* cardiac insufficiency

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Dosimetry of normal organs and tumors | through study completion, an average of 4 weeks
  The semiquantitative dosimetry will be performed based on SPECT/CT acquisitions after the first administration of 177Lu-LNC1011. The dose delivered to normal organs and tumors will be recorded.
Hematologic adverse events collection | through study completion, an average of 6 months
  Hematologic status were performed before and every 2 weeks after administration of radiopharmaceutical. Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0:Total white cell count less than 2.5 × 10^9/L,Platelet count less than 75 × 10^9/L
Liver and renal toxic events collection | through study completion, an average of 6 months
  Liver and renal function were performed before and 4 weeks after administration of radiopharmaceutical. Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0:Progressive deterioration of organ function (GFR <30 mL/min or creatinine > 2-fold upper limit of normal (ULN); liver enzymes > 5-fold ULN).

SECONDARY OUTCOMES:
PSA Response | through study completion, an average of 6 months
  The serum PSA response was documented semimonthly until 6 weeks after the administration of 177Lu-LNC1011. PSA response was classified as the following: partial response (PR) if PSA decrease ≥50%, progressive disease (PD) if PSA increase ≥ 25% and stable disease (SD) if PSA increase <25% or PSA decrease <50%.
Pharmacokinetics and dosimetry | Whole-body (WB) scans were performed at 2, 4, 24, 48, 72, 120, and 168 hours following intravenous administration of [177Lu]Lu-LNC1011
  Absorbed doses were measured in the brain, salivary glands, thyroid, cardiac content, lungs, liver, kidneys, spleen, pancreas, L2-L4 lumbar vertebrae, gastric content, and bladder content.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China